CLINICAL TRIAL: NCT00433992
Title: Effects of Thymidine Sparing Regimens on Mitochondrial Metabolism and Adipocyte Apoptosis
Brief Title: Metabolic Effects of Non-Thymidine Analogue Anti-HIV Medications
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Grace McComsey, Grace McComsey, MD, Case School of Medicine, National Institute of Allergy and Infectious Diseases (NIAID)
Other Study IDs: 1R01AI065348-01A2 (NIH)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections
Keywords: Mitochondria; Fat apoptosis; Lipoatrophy; Lipodystrophy; Thymidine; Treatment experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ABC/3TC: HIV-infected subjects were given Abacavir-Lamuvidine
- TDF/FTC: HIV-infected patients were given tenofovir DF-emtricitabine

SUMMARY:
The purpose of this study is to observe the effects of certain anti-HIV medications on mitochondrial activity and fat cell death. This study will enroll participants from another study, ACTG A5202, who are on treatment regimens that do not include zidovudine, stavudine, or other thymidine-containing anti-HIV medications.

DETAILED DESCRIPTION:
The main objective of this study is to observe the effects of anti-HIV medication lacking thymidine on mitochondrial metabolism and adipocyte apoptosis (fat cell death). Changes in mitochondrial metabolism and increases in adipocyte apoptosis are associated with lipoatrophy. Lipoatrophy is a common condition characterized by loss of subcutaneous fat and can be caused by many anti-HIV medications. This study will examine the metabolic consequences of the use of thymidine analogue-sparing treatment regimens.

This study will evaluate HIV infected patients who are enrolled in ACTG A5202, starting their first nucleoside reverse transcriptase inhibitor (NRTI)-containing regimen. This regimen will include either tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) or abacavir/lamivudine (ABC/3TC), which are thymidine-sparing regimens. The changes in mitochondrial activity and fat cell death will be compared between participants taking thymidine-sparing regimens (TDF/FTC or ABC/3TC) and thymidine-containing regimens.

This study will last for 96 weeks, with two study visits occurring at entry and another visit at Week 96. During each visit, a dual energy x-ray absorptiometry (DEXA) scan and blood collection will occur, and a fat biopsy will be performed in the lower abdomen under local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Enrolling in ACTG A5202 and its metabolic substudy ACTG A5224

Exclusion Criteria:

* Bleeding problems
* Cannot undergo fat biopsies
* Require aspirin anytime in the 7-day period prior to each biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who are enrolled in ACTG A5202, starting their first nucleoside reverse transcriptase inhibitor (NRTI)-containing regimen
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — Case School of Medicine
Locations (1):
- Case School of Medicine, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information on ACTG A5202 and ACTG 5224 — http://www.clinicaltrials.gov/ct/show/NCT00118898

RESULTS

PARTICIPANT FLOW:
Groups:
- ABC/3TC: HIV-infected subjects taking abacavir-lamivudine (ABC/3TC)
- TDF/FTC: HIV-infected subjects taking tenofovir DF-emtricitabine (TDF/FTC) with efavirenz (EFV) or atazanavir-lamivudine (ATV-r)
Period: Overall Study
Arm/Group | ABC/3TC | TDF/FTC
Started | 28 | 28
Completed | 19 | 20
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABC/3TC | TDF/FTC | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Mitochondrial Activity
Description: mtDNA content in adipose tissue was measured by quantitative real-time polymerase chain-reaction.
Time Frame: Entry, Week 96
Measure: Median (Inter-Quartile Range); unit: copies/cell
Groups:
- ABC/3TC+EFV: HIV-infected subjects taking abacavir-lamivudine (ABC/3TC) with Efavirenz at baseline
- TDF/FTC+EFV: HIV-infected subjects taking tenofovir DF-emtricitabine (TDF/FTC) with Efavirenz at baseline
- ATV/r +TDF/FTC: HIV infected subjects taking atazanavir-ritonavir with tenofovir DF-emtricitabine at baseline
- ATV/r +ABC/3TC: HIV-infected subjects taking atazanavir-ritonavir with abacavir-lamivudine at baseline
Arm/Group | ABC/3TC+EFV | TDF/FTC+EFV | ATV/r +TDF/FTC | ATV/r +ABC/3TC
Number analyzed (Participants) | 15 | 13 | 15 | 13
copies/cell | 1250 [998 to 1886] | 1312 [920 to 1609] | 1150 [721 to 1423] | 1125 [1049 to 1588]

2. Secondary Outcome: Change in Fat Apoptosis
Description: Changes in limb fat from 0 to 48 weeks measured with whole-body dual-energy x-ray absorptiometry
Time Frame: Entry, Week 48
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | ABC/3TC | TDF/FTC
Number analyzed (Participants) | 19 | 20
g | 906 [-349 to 1900] | 1479 [353 to 3032]

ADVERSE EVENTS:
Time Frame: the adverse event data was collected over the duration of the study of 96 weeks
Arm/Group | ABC/3TC | TDF/FTC
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/28
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABC/3TC (N=28) | TDF/FTC (N=28)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations included small sample size and premature study discontinuation before week 96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No